CLINICAL TRIAL: NCT01835093
Title: Tipepidine for ADHD
Brief Title: An Open Study of Tipepidine Hibenzate in Patients With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiba University (Other)
Responsible Party: Principal Investigator, Tsuyoshi Sasaki, Assistant Professor, Chiba University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G24061
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — tipepidine

ARMS (1):
- A single-arm study (Experimental)
  Interventions: Drug: Tipepidine Hibenzate

INTERVENTIONS:
Drug: Tipepidine Hibenzate

SUMMARY:
Accumulating evidence suggests a role of G protein-coupled inwardly-rectifying potassium (GIRK) channel in the pathology of excitement of nerve, and the medicine with the action (like the Tipepidine Hibenzate) is expected as a new curative medicine of Attention Deficit / Hyperactivity Disorder (AD/HD).

The purpose of this research is to confirm the effect by carrying out the additional dosage of the Tipepidine Hibenzate to the AD/HD patients.

If suggestion is obtained by this research about the effect on AD/HD of Tipepidine Hibenzate, it can contribute to development of the medical treatment of AD/HD.

ELIGIBILITY:
[Inclusion Criteria]

1. Attention-Deficit/Hyperactivity Disorder (AD/HD) for DSM-IV TR criteria.
2. Patients are treated with Atomoxetine, Methylphenidate, atypical antipsychotic drugs (risperidone, olanzapine, quetiapine, perospirone, aripiprazole, blonanserin, paliperidone) or not treated.
3. Patients are stable for 4-weeks for medication.

[Exclusion Criteria]

1. Patients with a previous hypersensitivity to Tipepidine Hibenzate.
2. Patients treated with typical antipsychotics and selective norepinephrine reuptake inhibitor (NRI) except atomoxetine and stimulants except methylphenidate.
3. Pregnant or breast-feeding women

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
ADHD Rating Scale-IV (ADHD-RS) Japanese Version | Changes from baseline in ADHD-RS at 4-weeks
  The ADHD Rating Scale-IV obtains parent ratings regarding the frequency of each ADHD symptom based on DSM-IV criteria.
  The ADHD Rating Scale-IV is completed independently by the parent and scored by a clinician. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items).

SECONDARY OUTCOMES:
Cognition using DN-CAS (Das-Naglieri Cognitive Assessment System) Japanese Version | Change from baseline in the scores of battery at 4-weeks
  The DN-CAS is an assessment battery designed to evaluate cognitive processing. It was developed to integrate theoretical and applied areas of psychological knowledge using cognitive processing theory and tests designed to measure-Planning, Attention, Simultaneous, and Successive Processing (PASS)-in individuals ages 5-17.
  This assessment facilitates mental health professionals in the identification of Attention-Deficit/Hyperactivity Disorder, Traumatic Brain Injury, learning disabilities, Mental Retardation, and giftedness.

CONTACTS AND LOCATIONS:
Overall Officials: Masaomi Iyo, MD,PhD, Study Chair — Chairman, Department of Psychiatry, Chiba University Graduate School of Medicine
Locations (1):
- Department of Psychiatry, Chiba University School of Medicine, Chiba, Chuo-ku, Japan

REFERENCES:
- [Result] Sasaki T, Hashimoto K, Tachibana M, Kurata T, Okawada K, Ishikawa M, Kimura H, Komatsu H, Ishikawa M, Hasegawa T, Shiina A, Hashimoto T, Kanahara N, Shiraishi T, Iyo M. Tipepidine in children with attention deficit/hyperactivity disorder: a 4-week, open-label, preliminary study. Neuropsychiatr Dis Treat. 2014 Jan 24;10:147-51. doi: 10.2147/NDT.S58480. eCollection 2014. PMID 24493927